CLINICAL TRIAL: NCT07143877
Title: Prognostic Impacts of Lipid Profile and Body Mass Index in Adult Acute Myeloid Leukemia Patients Treated With Intensive Induction Chemotherapy
Brief Title: Prognostic Impacts of Lipid Profile and BMI in Adult AML
Acronym: AML/BMI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Sayed Mohammad Bakheet, Resident of internal medicine department, Assiut University
Other Study IDs: 04-2025-201323
Record Dates: First submitted 2025-08-15; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: AML (Acute Myeloid Leukemia); BMI; Lipid Profile; Induction Chemotherapy
Keywords: AML; BMI; Lipid profile; Adult; Induction chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 35 Days

SUMMARY:
The goal of this observational study is to evaluate the changes in lipid profile parameters (total cholesterol, triglycerides, HDL-C, and LDL-C) in adult AML patients before and after intensive induction chemotherapy. The main questions it aims to answer are:

* Are there correlations between metabolic changes (in lipid profile and BMI) and treatment outcomes, including remission status and incidence of chemotherapy-related complications?
* Can the baseline lipid profile and BMI serve as prognostic markers for response to induction chemotherapy.?

Participants will be observed before and after induction chemotherapy regarding their lipid profile, and BMI, observing any correlations between the different results with any complications, and with remission status.

DETAILED DESCRIPTION:
Acute Myeloid Leukemia is a heterogeneous hematological malignancy characterized by clonal proliferation and accumulation of immature myeloid cells in the bone marrow and peripheral blood. It predominantly affects adults and often requires aggressive treatment in the form of intensive induction chemotherapy, typically based on cytarabine and anthracyclines.

The metabolic state of patients with AML including their lipid profile and body mass index, can influence both the disease course and response to treatment. Chemotherapy and its associated complications-such as infections, inflammation, and nutritional deficiencies-may lead to profound alterations in lipid metabolism and body composition.

Dyslipidemia may also emerge as a side effect of supportive medications like corticosteroids or parenteral nutrition. BMI is a simple anthropometric indicator of nutritional and general health status. Both undernutrition and obesity have been linked to adverse outcomes in cancer patients, including increased treatment-related toxicity and inferior survival rates. Similarly, changes in lipid parameters-such as total cholesterol, triglycerides, HDL, and LDL-may reflect systemic inflammation or hepatic dysfunction during treatment.

Given the rising interest in the metabolic implications of chemotherapy, it becomes imperative to investigate how intensive treatment affects these parameters in AML patients. However, there is a paucity of local data, particularly in Egyptian settings such as Assiut University Hospitals, where nutritional profiles and healthcare practices may differ from global norms.

Studying the lipid profile and BMI before and after induction chemotherapy may help identify at-risk patients, guide supportive care, and contribute to personalized treatment planning. This research aims to bridge the gap by exploring these metabolic indicators in adult AML patients managed at the Hematology Department of Assiut University Hospitals.

Study tools include patients' demographics including (age, sex, residence, occupation and age at time of diagnosis), detailed clinical history and physical examination, recording of demographic data (age and gender) and disease characteristics (AML subtype). Documentation of weight and height to calculate BMI before and after induction chemotherapy. Metabolic confounders (e.g.DM and Thyroid diseases) could be ruled out by History and examination. Laboratory tests would include Complete lipid profile (total cholesterol, triglycerides, HDL-C and LDL-C) measured at baseline and after completion of induction therapy. Complete blood count (CBC), liver function tests (LFTs), renal function tests, bone marrow aspirate for AML diagnosis and monitoring, and medication received

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18yearsold) newly diagnosed with AML.
* Patients eligible for intensive induction chemotherapy.
* Patients who have given informed consent to participate in the study.

Exclusion Criteria:

* Patients with secondary or relapsed AML.
* Patients currently using lipid-lowering medications (e.g., statins).
* Patients with known endocrine or metabolic disorders affecting BMI or lipid profile (e.g., uncontrolled diabetes, hypothyroidism, Cushing's syndrome).
* Pregnant or lactating women.
* Patients unwilling or unable to complete the study protocol.
* Patients with M3 subtype of AML.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients(≥18yearsold) newly diagnosed with AML.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Changes in lipid profile | Pre-induction to post-induction (day 28-35).
  Observing changes of lipid profile (total cholesterol, triglycerides, HDL-C, LDL-C) measured at baseline and after completion of induction therapy
Changes in Body Mass Index | Pre-induction to post-induction (day 28-35)
  Observing changes of Body Mass Index (measured as weight in kilograms divided by squared height in meters) measured at baseline and after completion of induction therapy

SECONDARY OUTCOMES:
Association of lipid profile changes with treatment response | Pre-induction to post-induction (day 28-35).
  Observing association of lipid profile changes with treatment response (complete remission, partial response, failure), occurrence of treatment-related complications (e.g., infections, tumor lysis syndrome), and duration of hospitalization.
Association of Body Mass Index changes with treatment response | Pre-induction to post-induction (day 28-35)
  Observing association of Body Mass Index (measures as weight in kilograms divided by squared height in meters) changes with treatment response (complete remission, partial response, failure), occurrence of treatment-related complications (e.g., infections, tumor lysis syndrome), and duration of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad S Mohammad, MBBS, Principal Investigator — Assiut University
Locations (1):
- Assiut university Hospitals, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No